CLINICAL TRIAL: NCT00096512
Title: Phase II Evaluation of BAY 43-9006 (NSC-724772) in Patients With Recurrent or Metastatic Head and Neck Cancer
Brief Title: S0420, Sorafenib in Treating Patients With Recurrent or Metastatic Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03043; S0420; U10CA032102 (NIH); CDR0000393212 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-11-09; First posted 2004-11-10 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Metastatic Squamous Neck Cancer With Occult Primary Squamous Cell Carcinoma; Recurrent Metastatic Squamous Neck Cancer With Occult Primary; Recurrent Salivary Gland Cancer; Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Nasopharynx; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Recurrent Verrucous Carcinoma of the Larynx; Recurrent Verrucous Carcinoma of the Oral Cavity; Salivary Gland Squamous Cell Carcinoma; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IVA Salivary Gland Cancer; Stage IVA Squamous Cell Carcinoma of the Larynx; Stage IVA Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVA Squamous Cell Carcinoma of the Oropharynx; Stage IVA Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVA Verrucous Carcinoma of the Larynx; Stage IVA Verrucous Carcinoma of the Oral Cavity; Stage IVB Salivary Gland Cancer; Stage IVB Squamous Cell Carcinoma of the Larynx; Stage IVB Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVB Squamous Cell Carcinoma of the Oropharynx; Stage IVB Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVB Verrucous Carcinoma of the Larynx; Stage IVB Verrucous Carcinoma of the Oral Cavity; Stage IVC Salivary Gland Cancer; Stage IVC Squamous Cell Carcinoma of the Larynx; Stage IVC Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVC Squamous Cell Carcinoma of the Oropharynx; Stage IVC Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVC Verrucous Carcinoma of the Larynx; Stage IVC Verrucous Carcinoma of the Oral Cavity; Tongue Cancer; Untreated Metastatic Squamous Neck Cancer With Occult Primary
MeSH Terms: conditions — Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms | interventions — Sorafenib

ARMS (1):
- Treatment (sorafenib tosylate) (Experimental): Patients receive oral sorafenib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sorafenib tosylate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: sorafenib tosylate — Given orally
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Sorafenib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. It may also stop the growth of tumor cells by stopping blood flow to the tumor. This phase II trial is studying how well sorafenib works in treating patients with recurrent or metastatic head and neck cance

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the response probability (confirmed, complete and partial responses) in patients with metastatic head and neck cancer who are treated with BAY 43-9006.

II. To evaluate median progression-free survival and median overall survival. III. To evaluate the qualitative and quantitative toxicities of this regimen. IV. To investigate in a preliminary manner the effects of the agent on the Ras signal transduction pathway in tissue samples obtained prior to and after treatment.

OUTLINE: This is a multicenter study.

Patients receive oral sorafenib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year and then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued for this study within 3.3-8 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically proven squamous cell carcinoma of the head and neck region that is either metastatic at diagnosis or has persisted, metastasized or recurred following definitive surgery and/or radiation therapy and is not amenable to salvage surgical resection; selected patients who have relapsed following prior induction or adjuvant therapy are eligible; patients with newly diagnosed non-metastatic disease are not eligible
* Patients must be willing to submit archived tissue specimens for immunohistochemistry correlative studies; the tissue can be from either the primary or metastatic site
* Patients must not have received prior chemotherapy for the recurrent or newly diagnosed metastatic disease; patients who have received induction or adjuvant chemotherapy are eligible, provided that at least six months have elapsed since the last course of chemotherapy was administered; patients may have received only one induction or adjuvant regimen
* Prior radiation must have been completed at least 28 days prior to registration and all toxicities must have been resolved
* Surgery must have been completed at least 28 days prior to registration and all complications/adverse events must have been resolved
* Patients must have measurable disease; all measurable disease must be assessed within 28 days prior to registration; if the patient also has non-measurable disease, then non-measurable disease must be assessed within 42 days prior to registration; patients whose only measurable disease is within a previous radiation therapy port must demonstrate clearly progressive disease (in the opinion of the treating investigator) prior to registration
* Patients must not be planning to receive any other concurrent therapy (i.e. radiation, chemotherapy, immunotherapy, biological therapy or gene therapy) for squamous cell carcinoma of the head and neck (SCCHN) while they are on this study
* Patients must have a Zubrod performance status of 0 or 1
* Patients with active infection requiring systemic therapy are not eligible
* Patients with active or prior central nervous system (CNS) metastasis are not eligible
* Granulocyte count > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Serum creatinine < 2 x the institutional upper limit of normal
* Bilirubin =< 2 x the institutional upper limit of normal
* Alkaline phosphatase =< 2 x the institutional upper limit of normal
* SGOT or SGPT =< 2 x the institutional upper limit of normal
* Patients must not have psychological, familial, sociological, or geographical conditions that prevent medical follow-up and compliance with the protocol treatment
* Patients must not have a significant history of cardiac disease, e.g., uncontrolled hypertension, unstable angina, congestive-heart failure, and myocardial infarction within the last six months, or cardiac ventricular arrhythmias requiring medication
* Patients must either be able to take oral medication without crushing, dissolving or chewing tablets
* Patients must not have any evidence of bleeding diathesis
* Patients must not be on therapeutic anticoagulation
* No prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for five years
* Pregnant or nursing women may not participate in this trial; women/men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method
* If day 28 or 42 falls on a weekend or holiday, the limit may be extended to the next working day
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* At the time of patient registration, the treating institution's name and ID number must be provided to the Data Operations Center in Seattle in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered into the data base

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-10; Primary Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Response | Up to 3 years
Progression-free survival | From date of registration to date of first observation of progressive disease, death due to any cause, symptomatic deterioration, assessed up to 3 years
  A 95% confidence interval will be provided.
Overall survival | From date of registration to date of death due to any cause, assessed up to 3 years
  A 95% confidence interval will be provided.
Toxicities assessed using NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 | Up to 3 years
  A 95% confidence interval will be provided.
Effects of the agent on the Ras signal transduction pathway | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Williamson, Principal Investigator — SWOG Cancer Research Network
Locations (1):
- Southwest Oncology Group (SWOG) Research Base, San Antonio, Texas, United States